CLINICAL TRIAL: NCT01306942
Title: A Phase I/II Trial of Dasatinib in Combination With Trastuzumab and Paclitaxel in the First Line Treatment of Her2-Positive Metastatic Breast Cancer (MBC) Patients
Brief Title: Dasatinib In Combination With Trastuzumab And Paclitaxel In First Line Treatment Of Her2-Positive MBC Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Spanish Breast Cancer Research Group (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEICAM/2010-04; 2010-023304-27 (EudraCT Number)
Record Dates: First submitted 2011-02-24; First posted 2011-03-02 (Estimated); Results first posted 2019-09-09 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Metastatic Breast Cancer
Keywords: HER2 positive breast cancer; first line treatment; Dasatinib; SRC kinase; Trastuzumab resistance
MeSH Terms: conditions — Breast Neoplasms | interventions — Dasatinib; Trastuzumab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dasatinib + trastuzumab + paclitaxel (Experimental): Eligible patients will be enrolled and treated with 4-week cycles of trastuzumab 2 mg/kg IV weekly (following a loading dose of 4 mg/kg in cycle 1) and paclitaxel 80 mg/m2 weekly x 3 weeks followed by a rest period of 7 days. Dasatinib will be administered orally in two dose levels 100 and 140 mg once daily (QD) (a -1 dose level is included just in case dose de-escalation is needed). Treatment will be repeated on Day 1 of a 28-day cycle until radiographic or symptomatic progression or unacceptable toxicity occurs. Only in the phase I, the first cycle will last 38 days.
  Interventions: Drug: Dasatinib; Drug: Trastuzumab; Drug: Paclitaxel

INTERVENTIONS:
Drug: Dasatinib
  Other Names: Sprycel
Drug: Trastuzumab
  Other Names: Herceptin
Drug: Paclitaxel
  Other Names: Taxol

SUMMARY:
This is a single-arm, open-label, phase I/II study. In the phase I, patients with Human Epidermal Growth Factor Receptor 2 (HER2) positive MBC will be treated with paclitaxel, trastuzumab and increasing doses of dasatinib to determine the Maximum Tolerated Dose (MTD), Dose Limiting Toxicity (DLT) and Recommended Phase II Dose (RPD) of the combination. Once the RPD has been identified, 48 patients will be treated at that dose to evaluate the efficacy and safety of the combination in the phase II.

DETAILED DESCRIPTION:
Eligible patients will be enrolled and treated with 4-week cycles of trastuzumab 2 mg/kg IV weekly (following a loading dose of 4 mg/kg in cycle 1) and paclitaxel 80 mg/m2 weekly x 3 weeks followed by a rest period of 7 days. Dasatinib will be administered orally in two dose levels 100 and 140 mg once daily (a -1 dose level is included just in case dose de-escalation is needed). Treatment will be repeated on Day 1 of a 28-day cycle in all patients (both in the phase I as in the phase II) until radiographic or symptomatic progression or unacceptable toxicity occurs. Only in the phase I and in all patients included in every different dose level, the first cycle will last 38 days.

Primary Objective:

* To determine the maximum tolerated dose (MTD) and recommended phase II dose (RPD) of dasatinib in combination with fixed doses of trastuzumab and paclitaxel in HER2-positive MBC patients (Phase I).
* To determine the efficacy, measured by objective response rate (ORR) in HER2-positive MBC patients with measurable disease (Phase II).

Secondary Objective(s):

* To characterize the safety of the combination (in both phase I and phase II).
* To evaluate the Clinical Benefit Rate (CBR), Time to Progression (TTP), Progression Free Survival (PFS) and Response Duration (RD) (in the phase II).
* To evaluate the pharmacokinetics (PK) of the combination (in the phase I and selected patients in the phase II if necessary).
* To evaluate molecular characteristics that may be predictive of the activity (or lack of) and any correlation between the biological activity of the study treatment and the disease outcome.

Exploratory objective:

• To explore the correlation between the lymphocytosis and efficacy.

Sample Size:

Phase I: following the 3+3 rule, a minimum of 6 and a maximum of 12 patients will be recruited.

Phase II:Assuming 10% drop-out rate, 48 patients are required to enter the study.

The duration of the study, from first patient visit to last patient visit will be approximately 42 months.

ELIGIBILITY:
Inclusion Criteria:

1. Female with histologically confirmed breast cancer with documented metastasis.
2. Patients must have Human Epidermal Growth Factor Receptor 2 (HER2) overexpression by immunohistochemistry (3+, HercepTest®; DAKO) or a positive fluorescence in situ hybridization for HER2 amplification evaluated by central laboratory. It is recommended that a formalin-fixed paraffin embedded (FFPE) tumor tissue block from the metastatic site (or the primary tumor, if metastatic site not available) required for HER2 testing are provided.
3. Patients can have measurable or non measurable disease for the Phase I part. For the Phase II only patients with measurable disease defined per RECIST 1.1 will be included.
4. Signed Written Informed Consent.
5. Target Population:

   1. Patients with Performance Status (ECOG) of 0 or 1.
   2. Number of previous therapies allowed or previous therapies may have included:

      * Chemotherapy: no prior chemotherapy for MBC is permitted. Patients treated with adjuvant chemotherapy regimens based on taxanes are allowed to be included if they are fully recovered of any taxane associated toxicity and a minimum of 12 months have elapsed from the end of this therapy.
      * Hormonal Therapy: patients may have had prior hormonal therapy. All hormonal agents must be discontinued at least 3 weeks prior to study entry.
      * Radiation Therapy: patients may have had prior radiation therapy that has not exceeded 25% of the bone marrow reserve. A minimum of 21 days must have elapsed between the last dose of radiation and registration into the study. Patients must have recovered from any acute toxic effects from radiation prior to registration. Lesions that have been irradiated cannot be included as sites of measurable disease for the phase II unless clear tumor progression, according to RECIST criteria, has been documented in these lesions since the end of radiation therapy.
      * Previous Surgery: previous surgery is permitted provided that wound healing has occurred.
      * Anti-HER2 Therapies: no prior anti-HER2 therapy for MBC is permitted. Patients treated with adjuvant anti-HER2 therapies (including but not limited to trastuzumab and lapatinib) are allowed to be included if a minimum of 12 months have elapsed from the end of this therapy.
   3. Adequate Organ Function (...).
   4. Ability to take oral medication (dasatinib must be swallowed whole).
   5. Concomitant Medications

   i) Patient agrees to discontinue St. Johns Wort while receiving dasatinib therapy (discontinue St. Johns Wort at least 5 days before starting dasatinib) ii) Biphosphonates must not be initiated within 28 days prior to study therapy
6. Age and sex:

   f) Patient, age 18 years old. g) Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for at least 4 weeks after the last dose of study drug to minimize the risk of pregnancy. (...)

Exclusion Criteria:

1. Sex and reproductive status:

   1. WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for at least 4 weeks after the last dose of study drug
   2. Women who are pregnant or breastfeeding.
   3. Women with a positive pregnancy test
2. Target Disease Exceptions:

   a) Central nervous system (CNS) metastases which are not well controlled. Eligible patients must be asymptomatic, cannot be receiving steroids or anticancer treatment, and must be enrolled at least 1 month after the end of the radiotherapy treatment
3. Medical History and Concurrent Diseases

   1. No malignancy [other than the one treated in this study] which required radiotherapy or systemic treatment within the past 5 years.
   2. Concurrent medical condition which may increase the risk of toxicity, including: Pleural or pericardial effusion of any grade.
   3. Cardiac Symptoms; any of the following should be considered for exclusion:

   i) Uncontrolled angina, congestive heart failure or myocardial infarction (MI) within (6 months) ii). Patients with intercurrent cardiac dysfunction or left ventricular ejection fraction (LVEF) < 50%.

   iii) Diagnosed congenital long QT syndrome. iv) Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes).

   v) Prolonged corrected QT (QTc) interval on pre-entry electrocardiogram (450 msec).

   vi) Patients with hypokalemia or hypomagnesemia if it cannot be corrected prior to dasatinib administration.

   d) History of significant bleeding disorder unrelated to cancer, including: i) Diagnosed congenital bleeding disorders (e.g., von Willebrand's disease). ii) Diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies).

   iii) Ongoing or recent (≤ 3 months) significant gastrointestinal bleeding.
4. Allergies and Adverse Drug Reactions

   a) Patients with known allergy to any of the study drugs or their components.
5. Prohibited Treatments and/or Therapies

   a) Category I drugs that are generally accepted to have a risk of causing Torsades de Pointes including: (Patients must discontinue drug 7 days prior to starting dasatinib) i) quinidine, procainamide, disopyramide ii) amiodarone, sotalol, ibutilide, dofetilide iii) erythromycin, clarithromycin iv) chlorpromazine, haloperidol, mesoridazine, thioridazine, pimozide v) cisapride, bepridil, droperidol, methadone, arsenic, chloroquine, domperidone, halofantrine, levomethadyl, pentamidine, sparfloxacin, lidoflazine.

   b) Concurrent anti-cancer therapy c) Potent CYP3A4 inhibitors
6. Other exclusion criteria:

   1. Patients who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness.
   2. Patients with active or uncontrolled infections or with serious illnesses or medical conditions that would not permit the patient to be managed according to the protocol.
   3. Patients unable or unwilling to give written informed consent prior to study participation.
   4. Pre-existent motor or sensory neurotoxicity of severity ≥ grade 2 according to NCI common toxicity criteria (version 4.03).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2019-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Complejo Hospitalario Universitario de Albacete
Locations (8):
- Spain (8):
  - Instituto Catalán de Oncología de Barcelona (Hospital Duran i Reynalds), L'Hospitalet de Llobregat, Barcelona
  - Hospital Alvaro Cunqueiro, Vigo, Pontevedra
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Clinic i Provincial, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Clínico Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen del Rocío, Seville
  - Instituto Valenciano de Oncología, Valencia

REFERENCES:
- [Result] Ocana A, Gil-Martin M, Antolin S, Atienza M, Montano A, Ribelles N, Urruticoechea A, Falcon A, Pernas S, Orlando J, Montero JC, Escudero MJ, Benito S, Caballero R, Carrasco E, Rojo F, Pandiella A, Ruiz-Borrego M. Efficacy and safety of dasatinib with trastuzumab and paclitaxel in first line HER2-positive metastatic breast cancer: results from the phase II GEICAM/2010-04 study. Breast Cancer Res Treat. 2019 Apr;174(3):693-701. doi: 10.1007/s10549-018-05100-z. Epub 2019 Jan 3. PMID 30607629
- [Result] Ocana A, Gil-Martin M, Martin M, Rojo F, Antolin S, Guerrero A, Trigo JM, Munoz M, Pandiella A, Diego NG, Bezares S, Caballero R, Carrasco E, Urruticoechea A. A phase I study of the SRC kinase inhibitor dasatinib with trastuzumab and paclitaxel as first line therapy for patients with HER2-overexpressing advanced breast cancer. GEICAM/2010-04 study. Oncotarget. 2017 Apr 14;8(42):73144-73153. doi: 10.18632/oncotarget.17113. eCollection 2017 Sep 22. PMID 29069857
- See also: Spanish Breast Cancer Research Group (GEICAM) is a Spanish Breast Cancer Research Group — http://www.geicam.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Ten patients were enrolled at the phase I receiving at least one cycle of the combination. Six patients were included at Dose Level (DL) 1 and four patients at DL 2. One patient at DL 1 and two patients at DL 2 had a DLT. Twenty-seven patients were included at the phase II.
Groups:
- Dasatinib 100mg + Trastuzumab 2mg/kg + Paclitaxel 80mg/m2: Cohort 1: Eligible patients were enrolled and treated with 4-week cycles of trastuzumab 2 mg/kg IV weekly (following a loading dose of 4 mg/kg in cycle 1) and paclitaxel 80 mg/m2 weekly x 3 weeks followed by a rest period of 7 days. Dasatinib 100mg was administered orally once daily (QD). Treatment was repeated on Day 1 of a 28-day cycle until radiographic or symptomatic progression or unacceptable toxicity occured. Only in the phase I, the first cycle lasted 38 days.
- Dasatinib 140mg + Trastuzumab 2mg/kg + Paclitaxel 80mg/m2: Cohort 2: Eligible patients were enrolled and treated with 4-week cycles of trastuzumab 2 mg/kg IV weekly (following a loading dose of 4 mg/kg in cycle 1) and paclitaxel 80 mg/m2 weekly x 3 weeks followed by a rest period of 7 days. Dasatinib 140mg was administered orally once daily (QD). Treatment was repeated on Day 1 of a 28-day cycle until radiographic or symptomatic progression or unacceptable toxicity occured. Only in the phase I, the first cycle lasted 38 days.
- Dasatinib 70mg + Trastuzumab 2mg/kg + Paclitaxel 80mg/m2: Cohort 3: Eligible patients were enrolled and treated with 4-week cycles of trastuzumab 2 mg/kg IV weekly (following a loading dose of 4 mg/kg in cycle 1) and paclitaxel 80 mg/m2 weekly x 3 weeks followed by a rest period of 7 days. Dasatinib 70mg was administered orally once daily (QD). Treatment was repeated on Day 1 of a 28-day cycle until radiographic or symptomatic progression or unacceptable toxicity occured. Only in the phase I, the first cycle lasted 38 days.
- PhaseII Dasatinib 100mg/Trastuzumab 2mg/kg/Paclitaxel 80mg/m2: Phase II with recommended Phase II Dose (RP2D) Dasatinib 100mg: Eligible patients were enrolled and treated with 4-week cycles of trastuzumab 2 mg/kg IV weekly (following a loading dose of 4 mg/kg in cycle 1) and paclitaxel 80 mg/m2 weekly x 3 weeks followed by a rest period of 7 days. Dasatinib 100mg was administered orally once daily (QD). Treatment was repeated on Day 1 of a 28-day cycle until radiographic or symptomatic progression or unacceptable toxicity occured. Two patients from phase I with measurable disease and RP2D were included in the phase II analyses.
Period: Phase I
Arm/Group | Dasatinib 100mg + Trastuzumab 2mg/kg + Paclitaxel 80mg/m2 | Dasatinib 140mg + Trastuzumab 2mg/kg + Paclitaxel 80mg/m2 | Dasatinib 70mg + Trastuzumab 2mg/kg + Paclitaxel 80mg/m2 | PhaseII Dasatinib 100mg/Trastuzumab 2mg/kg/Paclitaxel 80mg/m2
Started | 6 | 4 | 0 | 0
Completed | 1 | 1 | 0 | 0
Not Completed | 5 | 3 | 0 | 0
Not completed — Adverse Event | 2 | 2 | 0 | 0
Not completed — Physician Decision | 3 | 1 | 0 | 0
Period: Phase II
Arm/Group | Dasatinib 100mg + Trastuzumab 2mg/kg + Paclitaxel 80mg/m2 | Dasatinib 140mg + Trastuzumab 2mg/kg + Paclitaxel 80mg/m2 | Dasatinib 70mg + Trastuzumab 2mg/kg + Paclitaxel 80mg/m2 | PhaseII Dasatinib 100mg/Trastuzumab 2mg/kg/Paclitaxel 80mg/m2
Started | 2 (Two patients from phase I with measurable disease and RP2D were included in the phase II analyses.) | 0 (Dasatinib 140mg was not the RP2D, so these patients were not included in the phase II analyses.) | 0 | 27
Completed | 0 | 0 | 0 | 11
Not Completed | 2 | 0 | 0 | 16
Not completed — Adverse Event | 0 | 0 | 0 | 6
Not completed — Physician Decision | 2 | 0 | 0 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Not finished treatment | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Two patients from phase I with measurable disease and RP2D 100mg were included in the phase II analyses, and there is only one statistical analysis with this population of 29 patients (27 patients from phase II + 2 patients from phase I) for phase II.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dasatinib 100mg + Trastuzumab 2mg/kg + Paclitaxel 80mg/m2 | Dasatinib 140mg + Trastuzumab 2mg/kg + Paclitaxel 80mg/m2 | PhaseII Dasatinib 100mg/Trastuzumab 2mg/kg/Paclitaxel 80mg/m2 | Total
Number analyzed (Participants) | 6 | 4 | 29 | 39
Age, Continuous [Median (Full Range); unit: years] | 44.44 [35.35 to 81.26] | 49.43 [47.76 to 73.34] | 49.18 [31.82 to 81.37] | 48.48 [31.82 to 81.37]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 29 | 39
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 5 | 4 | 28 | 37
  Hispanic | 1 | 0 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Spain | 6 | 4 | 29 | 39
Menopausal Status [Count of Participants; unit: Participants]
  Postmenopausal | 2 | 2 | 17 | 21
  Premenopausal | 4 | 1 | 12 | 17
  Perimenopausal | 0 | 1 | 0 | 1
Eastern Cooperative Oncology Group (ECOG) status [Count of Participants; unit: Participants] — Measure Description: ECOG score runs from 0 to 5, with 0 denoting perfect health and 5 death.
  0 - Asymptomatic
  1. - Symptomatic but completely ambulatory
  2. - Symptomatic, <50% in bed during the day
  3. - Symptomatic, >50% in bed, but not bedbound
  4. - Bedbound
  5. - Death
  Participants
    ECOG 0 | 2 | 3 | 18 | 23
    ECOG 1 | 4 | 1 | 11 | 16
Hormonal Receptor [Count of Participants; unit: Participants]
  Estrogen Receptor: Positive | 5 | 2 | 22 | 29
  Estrogen Receptor: Negative | 1 | 2 | 7 | 10
  Progesterone Receptor: Positive | 4 | 1 | 13 | 18
  Progesterone Receptor: Negative | 2 | 3 | 16 | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicity (DLT) Within the First Cycle of Dasatinib in Combination With Trastuzumab and Paclitaxel (Phase I)
Description: DLT was defined as the occurrence of any of the following adverse events or abnormal laboratory value (graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.03), assessed as possibly, probably or definitively related to study drugs, occurring within the first cycle of study treatment: Need of any dose modification within the first cycle due to toxicity, grade 3 or 4 neutropenia complicated with fever ≥38.5° C or infection, grade 4 neutropenia (absolute neutrophil count (ANC)<0.5x1000000000/L) of at least 7 days duration, grade 3 thrombocytopenia complicated by hemorrhage, grade 4 thrombocytopenia, any grade 4 non-hematologic toxicity, grade 3 non-hematologic toxicities except nausea, vomiting, or diarrhea that can be controlled by appropriate medical intervention or prophylaxis, inability to resume dosing for cycle 2 at the current dose level within 14 days due to treatment related toxicity.
Time Frame: Up to cycle 1
Measure: Count of Participants; unit: Participants
Groups:
- Phase I: Dasatinib 100mg/Trastuzumab 2mg/kg/Paclitaxel 80mg/m2: Cohort 1: Eligible patients were enrolled and treated with 4-week cycles of trastuzumab 2 mg/kg IV weekly (following a loading dose of 4 mg/kg in cycle 1) and paclitaxel 80 mg/m2 weekly x 3 weeks followed by a rest period of 7 days. Dasatinib 100mg was administered orally once daily (QD). Treatment was repeated on Day 1 of a 28-day cycle until radiographic or symptomatic progression or unacceptable toxicity occured. Only in the phase I, the first cycle lasted 38 days.
- Phase I: Dasatinib 140mg/Trastuzumab 2mg/kg/Paclitaxel 80mg/m2: Cohort 2: Eligible patients were enrolled and treated with 4-week cycles of trastuzumab 2 mg/kg IV weekly (following a loading dose of 4 mg/kg in cycle 1) and paclitaxel 80 mg/m2 weekly x 3 weeks followed by a rest period of 7 days. Dasatinib 140mg was administered orally once daily (QD). Treatment was repeated on Day 1 of a 28-day cycle until radiographic or symptomatic progression or unacceptable toxicity occured. Only in the phase I, the first cycle lasted 38 days.
Arm/Group | Phase I: Dasatinib 100mg/Trastuzumab 2mg/kg/Paclitaxel 80mg/m2 | Phase I: Dasatinib 140mg/Trastuzumab 2mg/kg/Paclitaxel 80mg/m2
Number analyzed (Participants) | 6 | 4
Participants | 1 | 2

2. Primary Outcome: Maximum Tolerated Dose (MTD) of Dasatinib in Combination With Trastuzumab and Paclitaxel (Phase I)
Description: MTD is determined by testing increasing doses of dasatinib on dose escalation cohorts 3 to 6 patients per dose level. MTD reflects the highest dose tested in which a DLT is experienced by 0 out of 3 or 1 out of 6 patients among the dose levels
Time Frame: Up to cycle 1
Measure: Number; unit: mg
Groups:
- Phase I: Dasatinib + Trastuzumab + Paclitaxel: Eligible patients were enrolled and treated with 4-week cycles of trastuzumab 2 mg/kg IV weekly (following a loading dose of 4 mg/kg in cycle 1) and paclitaxel 80 mg/m2 weekly x 3 weeks followed by a rest period of 7 days. Dasatinib was administered orally in two dose levels 100 and 140 mg once daily (QD). Treatment was repeated on Day 1 of a 28-day cycle until radiographic or symptomatic progression or unacceptable toxicity occured. Only in the phase I, the first cycle lasted 38 days.
Arm/Group | Phase I: Dasatinib + Trastuzumab + Paclitaxel
Number analyzed (Participants) | 10
mg | 100

3. Primary Outcome: Recommended Phase II Dose (RP2D) of Dasatinib in Combination With Trastuzumab and Paclitaxel (Phase I).
Description: The RP2D was decided by the investigators taken into consideration the information obtained in the study and based on the MTD. To define the RP2D, information about toxicity observed during the full treatment were taken into consideration (relative dose intensity and toxicity observed).
Time Frame: Up to cycle 1
Measure: Number; unit: mg
Arm/Group | Phase I: Dasatinib + Trastuzumab + Paclitaxel
Number analyzed (Participants) | 10
mg | 100

4. Primary Outcome: Objective Response Rate (ORR)
Description: Tumor response was assessed using Response Evaluation Criteria In Solid Tumors Criteria (RECIST 1.1) criteria. ORR is defined as the percentage of patients with a Complete Response (CR) or Partial Response (PR) out of the patients who had measurable disease at baseline. Per RECIST, Complete Response (CR) is defined as the disappearance of all target lesions; Partial Response (PR) is defined as an >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Through study treatment, an average of 24 months
Measure: Count of Participants; unit: Participants
Groups:
- Phase II:Dasatinib 100mg/Trastuzumab 2mg/kg/Paclitaxel 80mg/m2: Phase II with recommended Phase II Dose (RP2D) Dasatinib 100mg: Eligible patients were enrolled and treated with 4-week cycles of trastuzumab 2 mg/kg IV weekly (following a loading dose of 4 mg/kg in cycle 1) and paclitaxel 80 mg/m2 weekly x 3 weeks followed by a rest period of 7 days. Dasatinib 100mg was administered orally once daily (QD). Treatment was repeated on Day 1 of a 28-day cycle until radiographic or symptomatic progression or unacceptable toxicity occured. Two patients from phase I with measurable disease and RP2D were included in the phase II analyses.
Arm/Group | Phase II:Dasatinib 100mg/Trastuzumab 2mg/kg/Paclitaxel 80mg/m2
Number analyzed (Participants) | 29
Participants | 23

5. Secondary Outcome: The Number of Participants Who Experienced Adverse Events (AE)
Description: Safety was assessed by standard clinical (blood pressure, pulse and body temperature, electrocardiogram (ECG), left ventricular ejection fraction (LVEF)) and laboratory tests (hematology: hemoglobin, platelet count, red blood cells (RBC), white blood cells (WBC) with differential (neutrophils) and absolute lymphocyte count, and serum chemistry: alkaline phosphatase, alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin, creatinine, sodium, potassium, magnesium, phosphate and calcium). Adverse events grade were defined by the NCI CTCAE v 4.03.
Time Frame: Through study treatment, an average of 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Dasatinib 100mg + Trastuzumab 2mg/kg + Paclitaxel 80mg/m2 | Dasatinib 140mg + Trastuzumab 2mg/kg + Paclitaxel 80mg/m2 | PhaseII Dasatinib 100mg/Trastuzumab 2mg/kg/Paclitaxel 80mg/m2
Number analyzed (Participants) | 6 | 4 | 29
Participants | 6 | 4 | 29

6. Secondary Outcome: To Evaluate the Clinical Benefit Rate (CBR)
Description: Tumor response was assessed using Response Evaluation Criteria In Solid Tumors Criteria (RECIST 1.1) criteria. CBR is defined as the percentage of patients with a Complete Response (CR) or Partial Response (PR) plus stable disease lasting at least 6 months out of the efficacy population. Per RECIST, CR is defined as the disappearance of all target lesions; PR is defined as an >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Through study treatment, an average of 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II:Dasatinib 100mg/Trastuzumab 2mg/kg/Paclitaxel 80mg/m2
Number analyzed (Participants) | 29
Participants | 24

7. Secondary Outcome: Time to Progression (TTP)
Description: TTP is defined as the time from the date of the first dose to the first date of objectively determined progressive disease. For patients not known to have objectively-determined progressive disease, TTP will be censored at the date of the last objective progression-free assessment. For patients who receive subsequent systemic anticancer therapy (after discontinuation from the study treatment) prior to objective disease progression, TTP will be censored at the date of last objective progression-free assessment prior to the initiation of post-discontinuation systemic anticancer therapy.
Time Frame: Through study treatment, an average of 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II:Dasatinib 100mg/Trastuzumab 2mg/kg/Paclitaxel 80mg/m2
Number analyzed (Participants) | 29
months | 23.9 [14.9 to NA] — The upper limit of the Confidence Interval (CI) was censored due to upper limit has not been reached.

8. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from the date of the first dose to the first date of objectively determined progressive disease or death from any cause. For patients not known to have died as of the data cut-off date and who do not have objectively-determined progressive disease, PFS will be censored at the date of the last objective progression-free assessment. For patients who receive subsequent systemic anticancer therapy (after discontinuation from the study treatment) prior to objective disease progression or death, PFS will be censored at the date of last objective progression-free assessment prior to the initiation of post-discontinuation systemic anticancer therapy.
Time Frame: Through study treatment, an average of 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II:Dasatinib 100mg/Trastuzumab 2mg/kg/Paclitaxel 80mg/m2
Number analyzed (Participants) | 29
months | 23.9 [10.3 to NA] — The upper limit of the Confidence Interval (CI) was censored due to upper limit has not been reached.

9. Secondary Outcome: Response Duration (RD)
Description: Tumor response was assessed using Response Evaluation Criteria In Solid Tumors Criteria (RECIST 1.1) criteria. RD is defined as the time from the date when the measurement criteria are met for complete response (CR) or partial response (PR) (whichever status is recorded first) until the date of first observation of disease progression or death occurred. Per RECIST, CR is defined as the disappearance of all target lesions; PR is defined as an >=30% decrease in the sum of the longest diameter of target lesions. For responding patients not known to have died as of the data cut-off date and who do not have progression, RD will be censored at the date of last visit with adequate assessment. For responding patients who receive subsequent anticancer therapy (after discontinuation from the study treatment) prior to progression, RD will be censored at the date of last visit with adequate assessment prior to the initiation of post-discontinuation anticancer therapy.
Time Frame: Through study treatment, an average of 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II:Dasatinib 100mg/Trastuzumab 2mg/kg/Paclitaxel 80mg/m2
Number analyzed (Participants) | 23
months | 18.4 [7.4 to NA] — The upper limit of the Confidence Interval (CI) was censored due to upper limit has not been reached.

10. Secondary Outcome: Dasatinib Maximun Plasma Concentration (Cmax) Value (Pharmacokinetics (PK) Phase I)
Description: To assess the influence of the concomitant administration of paclitaxel and trastuzumab on dasatinib PKs, we compared dasatinib exposures alone (first PK occasion: day 2 of cycle 1) or combined (second PK occasion: day 18 on cycle 1).
  The mean profiles of dasatinib plasma concentrations were determined by dose and PK occasion.
Time Frame: Cycle 1 day 2 and day 18
Population: Two participant samples for cycle 1 day 18 could not be obtained.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase I: Dasatinib 100mg/Trastuzumab 2mg/kg/Paclitaxel 80mg/m2 | Phase I: Dasatinib 140mg/Trastuzumab 2mg/kg/Paclitaxel 80mg/m2
Number analyzed (Participants) | 6 | 3
ng/mL
  Day 2 Dasatinib alone | 191.0 (92.1) | 422.3 (56.4)
  Day 18 Dasatinib in combination P and T: number analyzed (Participants) | 4 | 3
  Day 18 Dasatinib in combination P and T | 78.4 (51.1) | 314.4 (153.6)

11. Secondary Outcome: Dasatinib Area Under the Plasma Concentration-time Curve (AUC) Value (Pharmacokinetics (PK) Phase I)
Description: To assess the influence of the concomitant administration of paclitaxel and trastuzumab on dasatinib PKs, we compared dasatinib exposures alone (first PK occasion: day 2 of cycle 1) or combined (second PK occasion: day 18 on cycle 1).
  The area under the plasma concentration-time curve from time zero to 8 hours post dose (AUC0-8) were calculated in all treated patients, as the dasatinib plasmatic half-life is very short and concentrations at 24 hours post dose could only be quantified in some patients.
Time Frame: Cycle 1 day 2 and day 18
Population: Two participant samples for cycle 1 day 18 could not be obtained.
Measure: Mean (Standard Deviation); unit: ng·h/mL
Arm/Group | Phase I: Dasatinib 100mg/Trastuzumab 2mg/kg/Paclitaxel 80mg/m2 | Phase I: Dasatinib 140mg/Trastuzumab 2mg/kg/Paclitaxel 80mg/m2
Number analyzed (Participants) | 6 | 3
ng·h/mL
  Day 2 Dasatinib alone | 530.6 (237.1) | 1159.2 (128.3)
  Day 18 Dasatinib in combination P and T: number analyzed (Participants) | 4 | 3
  Day 18 Dasatinib in combination P and T | 248.1 (156.7) | 1047.3 (682.8)

12. Secondary Outcome: Phosphorylated SRC (p-SRC) Protein Expression Change in Peripheral Blood Mononuclear Cells After 8 Hours of Treatment (Phase II)
Description: Sequential peripheral blood mononuclear cells (PBMCs) on Cycle 1 Day 1 before treatment and 8 hours (h) after treatment (0h and 8h) were assessed to explore changes in the expression of p-SRC proteins measured by enzyme-linked immunosorbent assay (ELISA). For ELISA analyses, a duplicate of 100 µg of the extract was used to detect p-SRC (Tyr416). ELISA is a plate-based assay technique designed for detecting and quantifying proteins. The instrumentation used for protein signal-detection is an absorbance spectrophotometer (AS), which measures Absorbance (A). A is the quantity of light absorbed by a sample. As different compounds absorb light at different wavelengths, an AS can be used to distinguish compounds by analyzing the pattern of wavelengths absorbed by a given sample. Additionally, the amount of light absorbed is directly proportional to the concentration of absorbing compounds in that sample, so an AS can also be used to determine concentrations of compounds in the sample.
Time Frame: Cycle 1 day 1 at 0 hours and at 8 hours
Measure: Mean (Standard Deviation); unit: Absorbance 450 nm
Arm/Group | Phase II:Dasatinib 100mg/Trastuzumab 2mg/kg/Paclitaxel 80mg/m2
Number analyzed (Participants) | 16
Absorbance 450 nm | 0.36 (0.378)

13. Secondary Outcome: Phosphorylated AKT (p-AKT) Protein Expression Change in Peripheral Blood Mononuclear Cells After 8 Hours of Treatment (Phase II)
Description: Sequential peripheral blood mononuclear cells (PBMCs) on Cycle 1 Day 1 before treatment and 8 hours (h) after treatment (0h and 8h) were assessed to explore changes in the expression of p-AKT proteins measured by enzyme-linked immunosorbent assay (ELISA). For ELISA analyses, a duplicate of 100 µg of the extract was used to detect p-AKT (Ser473). ELISA is a plate-based assay technique designed for detecting and quantifying proteins. The instrumentation used for protein signal-detection is an absorbance spectrophotometer (AS), which measures Absorbance (A). A is the quantity of light absorbed by a sample. As different compounds absorb light at different wavelengths, an AS can be used to distinguish compounds by analyzing the pattern of wavelengths absorbed by a given sample. Additionally, the amount of light absorbed is directly proportional to the concentration of absorbing compounds in that sample, so an AS can also be used to determine concentrations of compounds in the sample.
Time Frame: Cycle 1 day 1 at 0 hours and at 8 hours
Measure: Mean (Standard Deviation); unit: Absorbance 450 nm
Arm/Group | Phase II:Dasatinib 100mg/Trastuzumab 2mg/kg/Paclitaxel 80mg/m2
Number analyzed (Participants) | 16
Absorbance 450 nm | 0.04 (0.09)

14. Secondary Outcome: Phosphorylation Status of Phosphorylated SRC (p-SRC) in Skin After Treatment (Phase I)
Description: p-SRC was analyzed in the skin biopsies taken at cycle 1 day 1 at 0 hours and 8 hours, cycle 1 day 4 and cycle 2 day 1, only in patients accepting to participate.
  A semi-quantitative H-score (or "histo" score) determined by the estimation of the percentage of tumour cells positively stained with low, medium, or high staining intensity. The final score is determined after applying a weighting factor to each estimate. The formula used is H-score = (low %) × 1 + (medium %) × 2 + (high %) × 3, and the results ranged from minimum 0 to maximum 300.
  Aim: to confirm the mechanism of action identified in preclinical models where the combination of dasatinib and trastuzumab show a statistically significant reduction in the phosphorylated levels of SRC.
Time Frame: Cycle 1 day 1 at 0 hours and at 8 hours, cycle 1 day 4 and cycle 2 day 1
Population: Skin biopsies could only be obtained in 5 participants at cycle 1 day 1 at 0 hours and 8 hours, cycle 1 day 4 and cycle 2 day 1.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Phase I: Dasatinib + Trastuzumab + Paclitaxel
Number analyzed (Participants) | 5
score on a scale
  H-score Cycle 1, day 1, 0 hours | 103 [90 to 116]
  H-score Cycle 1, day 1, 8 hours | 28 [10 to 46]
  H-score Cycle 1, day 4 | 14 [4 to 24]
  H-score Cycle 2, day 1 | 20 [8 to 32]

15. Secondary Outcome: Phosphorylation Status of Phosphorylated SRC (p-SRC) in Skin After Treatment (Phase II)
Description: p-SRC was analyzed in the skin biopsies taken at cycle 1 day 1 at 0 hours and 8 hours, only in patients accepting to participate.
  A semi-quantitative H-score (or "histo" score) determined by the estimation of the percentage of tumour cells positively stained with low, medium, or high staining intensity. The final score is determined after applying a weighting factor to each estimate. The formula used is H-score = (low %) × 1 + (medium %) × 2 + (high %) × 3, and the results ranged from minimum 0 to maximum 300.
  Aim: to confirm the mechanism of action identified in preclinical models where the combination of dasatinib and trastuzumab show a statistically significant reduction in the phosphorylated levels of SRC.
Time Frame: Cycle 1 day 1 at 0 hours and at 8 hours
Population: Skin biopsies could only be obtained in 6 participants at cycle 1 day 1 at 0 hours and 8 hours.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Phase II:Dasatinib 100mg/Trastuzumab 2mg/kg/Paclitaxel 80mg/m2
Number analyzed (Participants) | 6
score on a scale
  H-score 0 hours | 105 [83 to 127]
  H-score 8 hours | 27 [10 to 44]

16. Secondary Outcome: Phosphorylation Status of Phosphorylated AKT (p-AKT) in Skin After Treatment (Phase I)
Description: p-AKT was analyzed in the skin biopsies taken at cycle 1, day 1 at 0 hours and 8 hours, and cycle 2 day 1, only in patients accepting to participate.
  A semi-quantitative H-score (or "histo" score) determined by the estimation of the percentage of tumour cells positively stained with low, medium, or high staining intensity. The final score is determined after applying a weighting factor to each estimate. The formula used is H-score = (low %) × 1 + (medium %) × 2 + (high %) × 3, and the results ranged from minimum 0 to maximum 300.
  Aim: to confirm the mechanism of action identified in preclinical models where the combination of dasatinib and trastuzumab show a statistically significant reduction in the phosphorylated levels of AKT
Time Frame: Cycle 1 day 1 at 0 hours and at 8 hours and cycle 2 day 1
Population: Skin biopsies could only be obtained in 5 participants at cycle 1 day 1 at 0 hours and 8 hours and cycle 2 day 1.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Phase I: Dasatinib + Trastuzumab + Paclitaxel
Number analyzed (Participants) | 5
score on a scale
  H-score Cycle 1, day 1, 0 hours | 65 [31 to 99]
  H-score Cycle 1, day 1, 8 hours | 20 [10 to 30]
  H-score Cycle 1, day 4, 8 hours | 10 [10 to 10]
  H-score Cycle 2, day 1, 8 hours | 13 [8 to 18]

17. Secondary Outcome: Phosphorylation Status of Phosphorylated AKT (p-AKT) in Skin After Treatment (Phase II)
Description: p-AKT was analyzed in the skin biopsies taken at cycle 1, day 1 at 0 hours and 8 hours, only in patients accepting to participate.
  A semi-quantitative H-score (or "histo" score) determined by the estimation of the percentage of tumour cells positively stained with low, medium, or high staining intensity. The final score is determined after applying a weighting factor to each estimate. The formula used is H-score = (low %) × 1 + (medium %) × 2 + (high %) × 3, and the results ranged from minimum 0 to maximum 300.
  Aim: to confirm the mechanism of action identified in preclinical models where the combination of dasatinib and trastuzumab show a statistically significant reduction in the phosphorylated levels of AKT
Time Frame: Cycle 1 day 1 at 0 hours and at 8 hours
Population: Skin biopsies could only be obtained in 6 participants at cycle 1 day 1 at 0 hours and 8 hours.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Phase II:Dasatinib 100mg/Trastuzumab 2mg/kg/Paclitaxel 80mg/m2
Number analyzed (Participants) | 6
score on a scale
  H-score 0 hours | 70 [40 to 100]
  H-score 8 hours | 20 [10 to 30]

18. Secondary Outcome: Phosphorylation Status of Phosphorylated ERK (p-ERK) in Skin After Treatment (Phase I)
Description: p-ERK was analyzed in the skin biopsies taken at cycle 1 day 1 at 0 hours and 8 hours, cycle 1 day 4 at 8 hours, and cycle 2 day 1 at 8 hours, only in patients accepting to participate.
  A semi-quantitative H-score (or "histo" score) determined by the estimation of the percentage of tumour cells positively stained with low, medium, or high staining intensity. The final score is determined after applying a weighting factor to each estimate. The formula used is H-score = (low %) × 1 + (medium %) × 2 + (high %) × 3, and the results ranged from minimum 0 to maximum 300.
  Aim: to confirm the mechanism of action identified in preclinical models where the combination of dasatinib and trastuzumab show a statistically significant reduction in the phosphorylated levels of ERK
Time Frame: Cycle 1 day 1 at 0 hours and at 8 hours, cycle 1 day 4 at 8 hours and cycle 2 day 1 at 8 hours
Population: Skin biopsies could only be obtained in 5 participants at cycle 1 day 1 at 0 hours and 8 hours, cycle 1 day 4 at 8 hours and cycle 2 day 1 at 8 hours.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Phase I: Dasatinib + Trastuzumab + Paclitaxel
Number analyzed (Participants) | 5
score on a scale
  H-score Cycle 1, day 1, 0 hours | 63 [50 to 76]
  H-score Cycle 1, day 1, 8 hours | 20 [11 to 29]
  H-score Cycle 1, day 4, 8 hours | 14 [4 to 24]
  H-score Cycle 2, day 1, 8 hours | 11 [0 to 24]

19. Secondary Outcome: Phosphorylation Status of Phosphorylated ERK (p-ERK) in Skin After Treatment (Phase II)
Description: Phosphorylated extracellular signal-regulated kinases (p-ERK) 1 and 2 expression were analyzed in the skin biopsies taken at the cycle 1 day 1 at 0 hours and 8 hours, only in patients accepting to participate.
  A semi-quantitative H-score (or "histo" score) determined by the estimation of the percentage of tumour cells positively stained with low, medium, or high staining intensity. The final score is determined after applying a weighting factor to each estimate. The formula used is H-score = (low %) × 1 + (medium %) × 2 + (high %) × 3, and the results ranged from minimum 0 to maximum 300.
  Aim: to confirm the mechanism of action identified in preclinical models where the combination of dasatinib and trastuzumab show a statistically significant reduction in the phosphorylated levels of ERK
Time Frame: Cycle 1 day 1 at 0 hours and at 8 hours
Population: Skin biopsies could only be obtained in 6 participants at cycle 1 day 1 at 0 hours and 8 hours.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Phase II:Dasatinib 100mg/Trastuzumab 2mg/kg/Paclitaxel 80mg/m2
Number analyzed (Participants) | 6
score on a scale
  H-score 0 hours | 60 [49 to 71]
  H-score 8 hours | 16 [6 to 26]

20. Secondary Outcome: Number of Participants With Correlation Between Lymphocytosis and Efficacy.
Description: Efficacy (ORR, CBR, TTP, RD and PFS) was assessed using Response Evaluation Criteria In Solid Tumors Criteria (RECIST 1.1) criteria, and were correlated Lymphocytes, that were measured in the weekly hematology analyses performed within the first cycle.
Time Frame: Cycle 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dasatinib 100mg + Trastuzumab 2mg/kg + Paclitaxel 80mg/m2 | Dasatinib 140mg + Trastuzumab 2mg/kg + Paclitaxel 80mg/m2 | PhaseII Dasatinib 100mg/Trastuzumab 2mg/kg/Paclitaxel 80mg/m2
Number analyzed (Participants) | 6 | 4 | 29
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Through study treatment, an average of 12 months
Description: AE were reported after Informed Consent Document (ICD) and before study drugs until approximately 30 days following the discontinuation os study treatment.
Arm/Group | Dasatinib 100mg + Trastuzumab 2mg/kg + Paclitaxel 80mg/m2 | Dasatinib 140mg + Trastuzumab 2mg/kg + Paclitaxel 80mg/m2 | PhaseII Dasatinib 100mg/Trastuzumab 2mg/kg/Paclitaxel 80mg/m2
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/4 | 1/29
Serious Adverse Events (participants affected / at risk) | 1/6 | 2/4 | 6/29
Other Adverse Events (participants affected / at risk) | 6/6 | 4/4 | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dasatinib 100mg + Trastuzumab 2mg/kg + Paclitaxel 80mg/m2 (N=6) | Dasatinib 140mg + Trastuzumab 2mg/kg + Paclitaxel 80mg/m2 (N=4) | PhaseII Dasatinib 100mg/Trastuzumab 2mg/kg/Paclitaxel 80mg/m2 (N=29)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Grade 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — Grade 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — Grade 3
Angina (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — Grade 2
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Grade 3. Patient took dasatinib 140mg from January 30, 2014 to March 14, 2014. No any additional AEs were observed due to this intake of higher dose of dasatinib.
Soft tissue and skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Grade 3
Catheter related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Grade 2
Sudden death (General disorders) | 0 (0) | 0 (0) | 1 (1) — Grade 5
Febrile syndrome respiratory focus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — Grade 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dasatinib 100mg + Trastuzumab 2mg/kg + Paclitaxel 80mg/m2 (N=6) | Dasatinib 140mg + Trastuzumab 2mg/kg + Paclitaxel 80mg/m2 (N=4) | PhaseII Dasatinib 100mg/Trastuzumab 2mg/kg/Paclitaxel 80mg/m2 (N=29)
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 — Grade 3
Aspartate aminotransferase increased (Investigations) | 1 | 0 (0) | 0 — Grade 3
Diarrhea (Gastrointestinal disorders) | 2 | 0 | 1 — Grade 3
Fatigue (General disorders) | 1 | 1 | 2 — Grade 3
Hypertension (Vascular disorders) | 1 | 0 | 2 — Grade 3
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1 | 2 — Grade 3
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 — Grade 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 — Grade 3
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 — Grade 3
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 — Grade 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 — Grade 3
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 — Grade 3
Ejection Fraction Decreased (Investigations) | 0 | 0 | 3 — Grade 3
Anemia (Blood and lymphatic system disorders) | 3 | 3 | 12 — Grade 2
Ejection Fraction Decreased (Investigations) | 1 | 0 | 7 — Grade 2
Neutrophil Count Decreased (Investigations) | 0 | 1 | 7 — Grade 2
Neutrophil Count Decreased (Investigations) | 0 | 0 | 2 — Grade 3
Neutrophil Count Decreased (Investigations) | 4 | 1 | 16 — Grade 1
Weight Gain (Investigations) | 1 | 0 | 7 — Grade 2
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 0 | 13 — Grade 2
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 1 | 7 — Grade 2
Fatigue (General disorders) | 3 | 0 | 18 — Grade 1
Fatigue (General disorders) | 0 | 3 | 5 — Grade 2
Anorexia (Metabolism and nutrition disorders) | 0 | 3 | 1 — Grade 2
Alanine Aminotransferase Increased (Investigations) | 4 | 3 | 17 — Grade 1
Aspartate Aminotransferase Increased (Investigations) | 3 | 4 | 20 — Grade 1
Red Blood Cells Count Decrease (Investigations) | 5 | 4 | 27 — Grade 1
Anemia (Blood and lymphatic system disorders) | 3 | 1 | 13 — Grade 1
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 13 — Grade 1
White Blood Cell Decreased (Investigations) | 3 | 2 | 12 — Grade 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1 — Grade 1
Lymphopenia (Investigations) | 2 | 3 | 1 — Grade 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 — Grade 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 5 — Grade 1
Fever (General disorders) | 1 | 2 | 4 — Grade 1
Hypertension (Vascular disorders) | 1 | 2 | 5 — Grade 1
Edema limbs (General disorders) | 1 | 2 | 3 — Grade 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 1 | 2 — Grade 1
Anorexia (Metabolism and nutrition disorders) | 4 | 0 | 6 — Grade 1
Alkaline phosphatase increased (Investigations) | 3 | 0 | 9 — Grade 1
Headache (Nervous system disorders) | 3 | 1 | 5 — Grade 1
Mucositis oral (Gastrointestinal disorders) | 3 | 1 | 8 — Grade 1
Nausea (Gastrointestinal disorders) | 3 | 0 | 7 — Grade 1
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 1 | 11 — Grade 1
Activated Partial Thromboplastin Time Prolonged (Investigations) | 1 | 0 | 6 — Grade 2
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0 | 8 — Grade 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less